CLINICAL TRIAL: NCT00598637
Title: Prospective Randomized Trial of Everolimus- and Zotarolimus-eluting Stents for Treatment of Unprotected Left Main Coronary Artery Disease: ISAR-LEFT-MAIN-2
Brief Title: Drug-eluting Stents to Treat Unprotected Coronary Left Main Disease
Acronym: LEFT-MAIN-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S02807
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Disease
Keywords: drug eluting stent; left main disease
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EES (Active Comparator): Everolimus-eluting stent (Xience)
  Interventions: Device: Everolimus-eluting stent (Xience)
- ZES (Experimental): Zotarolimus-eluting stent (Endeavor Resolute)
  Interventions: Device: Zotarolimus-eluting stent (Endeavor Resolute)

INTERVENTIONS:
Device: Everolimus-eluting stent (Xience) — stent is implanted due to randomization
  Other Names: Xience
  Arms: EES
Device: Zotarolimus-eluting stent (Endeavor Resolute) — stent is implanted due to randomization
  Other Names: Endeavor Resolute
  Arms: ZES

SUMMARY:
The purpose of this study is to evaluate the efficacy of two different drug-eluting stents (Everolimus and Zotarolimus-eluting) for treatment of unprotected left main coronary artery disease.

DETAILED DESCRIPTION:
Restenosis in the left main coronary artery may have severe consequences given the large proportion of the myocardium compromised in this condition, and, in several studies, it has been linked to the 6-month mortality after the index procedure. Drug-eluting stents have reduced the restenosis rate and the need for target vessel revascularization not only in simple lesion but also in high risk subsets of patients and lesions such as diabetics, long lesions or bifurcations. There are no data about their efficacy in left main coronary artery disease. Thus, the aim of this study is to investigate the performance of two different drug-eluting stents (Everolimus and Zotarolimus-eluting) in left main coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50 % stenosis located in unprotected LMCA who are unable to undergo CABG because of cardiac surgeons' refusal (poor surgical candidates) or their own unwillingness.
* Pretreatment with a loading dose of 600 mg clopidogrel.
* Informed, written consent by the patients or her/his legally-authorized representative for participation in the study.

Exclusion Criteria:

* Cardiogenic shock.
* ST-segment elevation acute myocardial infarction (ST-segment ≥ 0.1 mV elevation in ≥ 2 contiguous ECG leads persisting for at least 20 minutes) within 48 hours from symptom onset.
* In-stent restenosis.
* Malignancies or other comorbid conditions with life expectancy less than one year or that may result in protocol non-compliance.
* Prior coronary artery bypass surgery with revascularization of LAD and/or LCx.
* Planned staged PCI procedure within 30 days from index procedure or prior PCI within the last 30 days.
* An elective surgical procedure is planned that would necessitate interruption of clopidogrel during the first six months post enrollment.
* Known allergy to the study medications: aspirin, clopidogrel, UHF; sirolimus, paclitaxel; true anaphylaxis after prior exposure to contrast media.
* Pregnancy (present, suspected or planned).
* Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2007-12; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac event defined as a composite of death, myocardial infarction and target lesion revascularization. | 1 year follow-up

SECONDARY OUTCOMES:
Angiographic restenosis at follow-up coronary angiography. | 6-9 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum Muenchen; Julinda Mehill, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (4):
- Germany (3):
  - Bad Segeberger Kliniken, Bad Segeberg
  - Deutsches Herzzentrum Muenchen, Munich
  - First Medizinische Klinik, Klinikum rechts der Isar, Munich
- Azienda Ospedaliero Universitaria di Ferrara, Ferrara, Italy

REFERENCES:
- [Background] Park SJ, Hong MK, Lee CW, Kim JJ, Song JK, Kang DH, Park SW, Mintz GS. Elective stenting of unprotected left main coronary artery stenosis: effect of debulking before stenting and intravascular ultrasound guidance. J Am Coll Cardiol. 2001 Oct;38(4):1054-60. doi: 10.1016/s0735-1097(01)01491-7. PMID 11583882
- [Background] Park SJ, Park SW, Hong MK, Cheong SS, Lee CW, Kim JJ, Hong MK, Mintz GS, Leon MB. Stenting of unprotected left main coronary artery stenoses: immediate and late outcomes. J Am Coll Cardiol. 1998 Jan;31(1):37-42. doi: 10.1016/s0735-1097(97)00425-7. PMID 9426015
- [Derived] Cassese S, Kufner S, Xhepa E, Byrne RA, Kreutzer J, Ibrahim T, Tiroch K, Valgimigli M, Tolg R, Fusaro M, Schunkert H, Laugwitz KL, Mehilli J, Kastrati A. Three-year efficacy and safety of new- versus early-generation drug-eluting stents for unprotected left main coronary artery disease insights from the ISAR-LEFT MAIN and ISAR-LEFT MAIN 2 trials. Clin Res Cardiol. 2016 Jul;105(7):575-84. doi: 10.1007/s00392-015-0953-x. Epub 2015 Dec 22. PMID 26689707
- [Derived] Mehilli J, Richardt G, Valgimigli M, Schulz S, Singh A, Abdel-Wahab M, Tiroch K, Pache J, Hausleiter J, Byrne RA, Ott I, Ibrahim T, Fusaro M, Seyfarth M, Laugwitz KL, Massberg S, Kastrati A; ISAR-LEFT-MAIN 2 Study Investigators. Zotarolimus- versus everolimus-eluting stents for unprotected left main coronary artery disease. J Am Coll Cardiol. 2013 Dec 3;62(22):2075-82. doi: 10.1016/j.jacc.2013.07.044. Epub 2013 Aug 21. PMID 23973699